CLINICAL TRIAL: NCT00489814
Title: Prospective Evaluation of Quality of Life After Proton Therapy for Prostate Cancer
Brief Title: Study of Quality of Life for Prostate Proton Therapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0956
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostate Proton Therapy; Proton Radiation Therapy; Proton Radiotherapy; Quality of Life; QOL; Questionnaire
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients who are planned to undergo local proton radiotherapy for biopsy-proven, untreated, prostate adenocarcinoma.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires administered within 3 weeks before the beginning of the radiation treatment course, twice during radiation therapy, and upon completion of radiation therapy.
  Other Names: Survey

SUMMARY:
The goal of this research study is to collect information on the side effects of proton radiation therapy given for the treatment of prostate cancer as well as the effect of proton therapy on quality of life. Information on your treatment and how you react to the treatment will be collected. Researchers will use this information to try to understand how people tolerate proton radiation therapy for prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer tends to be better controlled with higher doses of radiation. These high doses may lead to more side effects. Standard radiation therapy uses x-rays, which are effective but may cause extra radiation dose to be given to tissues beyond the tumor, such as the rectum and bladder. Unlike x-rays, protons (small positively-charged particles) can deliver radiation dose to a specific target but then suddenly deliver much less dose beyond the target. This minimizes the dose to normal tissues and may lead to fewer side effects, even when high doses are delivered to the tumor.

If you agree to take part in this study, it will involve completing quality of life questionnaires before, during, and after proton therapy. You will be asked how you tolerated the proton therapy, what (if any) side effects you experienced, and how the treatment impacts the quality of your life. The questionnaires should each take about 15 minutes to complete. They may be done in person, by mail, or by phone.

You will complete the questionnaires before the proton therapy begins and during the last week of therapy. You will also repeat the questionnaires at 3, 6, 9, and 12 months after the proton therapy, every 6 months for the next 3 years, and every year for the next 6 years after that. If you are receiving hormone therapy, you will also be asked to fill out a questionnaire before or at the beginning of hormone therapy. During your radiation course, you will have a brief weekly clinic visit and assessed for any side effects during that visit as part of normal standard practice. Your information will be compiled with the information from other people who were treated similarly, to better understand the effects of prostate proton radiation therapy.

Throughout the course of your radiation therapy, you will have brief clinic visits once a week as part of your standard care. You will be checked for any side effects.

Your participation in the study will be over after you mail back the last questionnaire.

This is an investigational study. Up to 1084 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are planned to undergo local proton radiotherapy for biopsy-proven, untreated, prostate adenocarcinoma with Gleason scoring.
2. 1992 AJCC clinical stage T1-T3c on digital rectal exam.
3. PSA within 4 weeks of study entry.
4. Zubrod performance status of 0-1 with a life expectancy of at least 10 years.
5. Prior hormonal therapy allowed if began no more than three months prior to registration.
6. Patient must be able to adhere to follow-up schedule either personally or via mail or phone.
7. Patient must be able to speak, read and understand English.
8. Patient must give informed consent.

Exclusion Criteria:

1. Histology other than adenocarcinoma.
2. Evidence of distant or nodal metastasis.
3. Prior pelvic radiotherapy or chemotherapy.
4. Prior or planned radical prostate surgery.
5. Prior local therapy for prostate cancer.
6. Previous and/or concurrent malignancy unless disease free for >5 years. Basal cell and non-invasive squamous cell carcinoma of the skin will not exclude patient from eligibility.
7. History of inflammatory bowel disease (e.g. Crohn's disease or ulcerative colitis).
8. Patients with metallic devices in the hip/pelvis (e.g. hip prostheses) that may interfere with proton dosimetry will not be eligible.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants who are planned to undergo local proton radiotherapy for biopsy-proven, untreated, prostate adenocarcinoma.
Sampling Method: Probability Sample
Enrollment: 1125 (Actual)
Dates: Start 2006-05-24 (Actual); Primary Completion 2020-05-24 (Estimated); Study Completion 2020-05-24 (Estimated)

PRIMARY OUTCOMES:
To collect information on the side effects of proton radiation therapy given for the treatment of prostate cancer as well as the effect of proton therapy on quality of life. | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Seungtaek Choi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org